CLINICAL TRIAL: NCT04344210
Title: Impact of Tele-Interventions During the COVID-19 Pandemic on Glycemic Control and Attitude Toward the Disease in Patients With Diabetes Mellitus - A Randomized Clinical Trial
Brief Title: Impact of Tele-interventions During the COVID-19 Pandemic in Patients With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Janine Alessi, Master Student, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020241093
Record Dates: First submitted 2020-04-07; First posted 2020-04-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: COVID; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: COVID-19; Diabetes Mellitus; Glycemic control; Tele-Intervention; Mental well-being
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; COVID-19; Diabetes Mellitus; Psychological Well-Being | interventions — Mental Health

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in two groups: G1: participants will receive a tele-intervention by a case manager weekly to discuss topics related to diabetes management and mental well-being during the quarantine period ; G2: participants will receive the usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Intervention (Experimental): Participants will receive a tele-intervention by a case manager weekly to discuss topics related to diabetes management and mental well-being during the quarantine period
  Interventions: Behavioral: Tele-interventions related to diabetes management and mental well-being
- Usual Care (No Intervention): Participants will receive the usual care

INTERVENTIONS:
Behavioral: Tele-interventions related to diabetes management and mental well-being — Participants will receive a tele-intervention by a case manager weekly to discuss topics related to diabetes management and mental well-being during the quarantine period
  Arms: Tele-Intervention

SUMMARY:
INTRODUCTION In critical situations, such as the current COVID 19 pandemic, themes of fear, uncertainty and stigmatization are common and constitute barriers to appropriate medical and mental health interventions. These challenges, when faced by those who live with a chronic disease, such as diabetes mellitus (DM), can negatively influence quality of life and adherence to treatment, compromising the control of the disease.

OBJECTIVES The present study aims to investigate the effectiveness of a tele-intervention during the COVID-19 pandemic in improving glycemic control, lipid profile, blood pressure levels and parameters of medication adherence, mental well-being and sleep quality in patients with type 1 DM and type 2 DM.

METHODS A randomized clinical trial will be carried out with patients with a previous diagnosis of type 1 DM and type 2 DM, who are registered at the Hospital de Clínicas de Porto Alegre (HCPA). Inclusion criteria will be age greater than or equal to 18 years, collection of HbA1c in the HCPA laboratory in January, February or March 2020 and availability to receive weekly phone calls. Patients will be randomized, stratified by type of diabetes, in two groups: G1: participants will receive a tele-intervention by a case manager weekly to discuss topics related to diabetes management and mental well-being during the social distancing period ; G2: participants will receive the usual care. The primary outcome assessed will be the variation in HbA1c levels comparatively between groups, with or without a tele-guided strategy, after four months of social distancing (or as long as the recommendation of social distancing measures remains). Secondary outcomes will include experiencing confirmation of COVID-19 infection, variation in lipid profile, blood pressure levels and variation in parameters of emotional distress related to diabetes, eating disorders, medication adherence, symptoms minor psychiatric disorders and altered sleep patterns, which will be evaluated with specific and validated scales. According to the sample calculation, 150 patients will be included in the study (92 with type 2 DM and 58 with type 1 DM). Analysis by intention to treat will be performed separately for patients with type 1 DM and with type 2 DM.

SCHEDULE The proposed experiment will start immediately after approval of this project by the research ethics committee. The duration of the proposed intervention is 4 months (or as long as the recommendation of social distancing measures remains. This means that the study may be completed before or after that period, based on national recommendations for social distancing in Brazil), with a data analysis plan and publication of the results until September 2020.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus or type 2 diabetes mellitus;
* Age greater than or equal to 18 years;
* HbA1c assessed in January, February or March 2020;
* Availability to receive weekly phone calls

Exclusion Criteria:

* Any severe cognitive limitation that prevents the necessary interaction to carry out this study (advanced dementia, deafness, dysarthria, aphasia);
* Do not present a telephone record in an electronic medical record;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Variation in HbA1c levels | 4 months (or as long as the recommendation of social distancing measures remains)
  Variation in HbA1c levels comparatively between groups after the period of social distancing measures.

SECONDARY OUTCOMES:
COVID-19 infection | 4 months (or as long as the recommendation of social distancing measures remains)
  Confirmation of coronavirus infection by rapid test
Variation in lipid profile | 4 months (or as long as the recommendation of social distancing measures remains)
  Comparison of the lipid profile of the last year with the lipid profile after the intervention between the groups.
Variation in blood pressure levels | 4 months (or as long as the recommendation of social distancing measures remains)
  Comparison of the blood pressure level of the last consultation with the pressure after the intervention between the groups.
Comparison of emotional distress associated with the routine of living with diabetes after intervention between groups | 4 months (or as long as the recommendation of social distancing measures remains)
  Evaluation of emotional distress associated with the routine of living with diabetes - B-PAID (Brazilian Problem Areas In Diabetes Scale)
Comparison of eating disorders between groups | 4 months (or as long as the recommendation of social distancing measures remains)
  Evaluation of eating disorders - EAT - 26 SCALE (Teste de Atitudes Alimentares)
Comparison of adherence to the proposed clinical treatment between groups | 4 months (or as long as the recommendation of social distancing measures remains)
  Evaluation of adherence to the proposed clinical treatment - SCI R (Self-Care Inventory - revised)
Comparison of minor psychiatric disorders between groups | 4 months (or as long as the recommendation of social distancing measures remains)
  Evaluation of minor psychiatric disorders - SRQ 20 (Self Report Questionnaire)
Comparison of sleep pattern changes between groups | 4 months (or as long as the recommendation of social distancing measures remains)
  Evaluation of sleep pattern changes - MSQ (Mini Sleep Questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Franco DW, Alessi J, de Carvalho TR, Kobe GL, Oliveira GB, Knijnik CP, Amaral B, Becker AS, Schaan BD, Telo GH. The impact of a telehealth intervention on the metabolic profile of diabetes mellitus patients during the COVID-19 pandemic - A randomized clinical trial. Prim Care Diabetes. 2022 Dec;16(6):745-752. doi: 10.1016/j.pcd.2022.09.011. Epub 2022 Sep 30. PMID 36266163
- [Derived] Alessi J, Becker AS, Amaral B, de Oliveira GB, Franco DW, Knijnik CP, Kobe GL, de Brito A, de Carvalho TR, Telo GH, Schaan BD, Telo GH. Type 1 diabetes and the challenges of emotional support in crisis situations: results from a feasibility study of a multidisciplinary teleintervention. Sci Rep. 2022 May 20;12(1):8526. doi: 10.1038/s41598-022-12227-z. PMID 35595850
- [Derived] Alessi J, Becker AS, Amaral B, de Oliveira GB, Franco DW, Knijnik CP, Kobe GL, de Brito A, de Carvalho TR, Telo GH, Schaan BD, Telo GH. Type 1 diabetes and the challenges of emotional support in crisis situations: results from a randomized clinical trial of a multidisciplinary teleintervention. Sci Rep. 2022 Feb 23;12(1):3086. doi: 10.1038/s41598-022-07005-w. PMID 35197493 (Retraction: PMID 35277576 Sci Rep. 2022 Mar 11;12(1):4265)